CLINICAL TRIAL: NCT04389970
Title: Time Restricted Eating Outcomes in Multiple Sclerosis
Acronym: TREO_MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Brooks C. Wingo, PhD, Associate Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 300005334-001; P30DK056336 (NIH)
Record Dates: First submitted 2020-05-07; First posted 2020-05-15 (Actual); Results first posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Multiple Sclerosis; Diet, Healthy
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Time Restricted Feeding (Experimental): Participants will be asked to follow a time-restricted meal pattern (8:16 protocol)
  Interventions: Behavioral: Time Restricted Feeding

INTERVENTIONS:
Behavioral: Time Restricted Feeding — Participants will eat all food within an 8 hour window each day. They will only consume water or black coffee during the remaining 16 hours.

SUMMARY:
The purpose of this pilot study is to determine the preliminary efficacy, safety, and acceptability of time restricted feeding (TRF) among a sample of 12 adults with Relapsing-Remitting Multiple Sclerosis (RRMS). The specific aims of this study are: 1: To determine preliminary efficacy of TRF for reducing symptom burden, improving inflammatory markers, and reducing cardiometabolic risk among adults with RRMS. 2: To determine the safety and participant acceptability of TRF. Participants will be asked to consume all food during an 8-hour window each day and not eat for the remaining 16 hours. All participants will follow this eating pattern for 8 weeks.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic autoimmune disease characterized by demyelination and loss of axons in the central nervous system. Over the last decade there has been an influx of evidence demonstrating the impact of lifestyle risk factors on the progression of MS symptoms. Specifically, epidemiological studies report that poor diet is associated with increased risk of disability in adults with MS. Despite this evidence, little research has explored dietary interventions that may reduce symptom burden of MS. One dietary intervention that has shown particular promise in animal models of MS is intermittent fasting (IF), which is a dietary pattern characterized by cycles of eating and extended fasting. There are a number of protocols for IF, including time restricted feeding (TRF), in which all food is consumed during a limited window of time each day. Growing evidence demonstrates that IF reduces inflammation, improves immune function, and improves cardiometabolic risk in animal models of MS, however, little of this research has been translated into human trials. In addition to these physiological benefits, the investigators believe that TRF will provide a behavioral benefit, as it addresses barriers traditionally seen in dietary interventions by shifting the focus from restricting what participants eat, to focusing on meal timing.

The purpose of this pilot study is to determine the preliminary efficacy, safety, and acceptability of TRF in adults with MS. The specific aims of this study are: 1: To determine preliminary efficacy of TRF for reducing symptom burden, improving inflammatory markers, and reducing cardiometabolic risk among adults with RRMS. 2: To determine the safety and participant acceptability of TRF.

Twelve adults with relapsing-remitting MS will eat all meals within an 8 hour period each day. All participants will follow the assigned meal plan for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Relapsing Remitting MS (RRMS)
* BMI between 18-50 kg.m2
* If on disease-modifying medications, stable for 6 months
* If not on disease-modifying medication, no medication usage within previous 6 months
* Able to walk 25 ft. with or without assistance

Exclusion Criteria:

* Relapse within previous 30 days
* Actively engaged in a weight loss program or unwilling to follow assigned dietary timing pattern
* Regularly fasts >15 hours/day
* Pregnant or breastfeeding
* Current use of insulin or sulfonylurea agents

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brooks C Wingo, PhD, Principal Investigator — Univeristy of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Wingo BC, Rinker JR 2nd, Green K, Peterson CM. Feasibility and acceptability of time-restricted eating in a group of adults with multiple sclerosis. Front Neurol. 2023 Jan 12;13:1087126. doi: 10.3389/fneur.2022.1087126. eCollection 2022. PMID 36712417

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Time Restricted Feeding
Started | 12
Completed | 11
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Time Restricted Feeding
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Timed 25-foot Walk Speed
Description: Change in timed 25-foot walk test speed between baseline and 8 weeks. Speed calculated as ft per second, and change calculated as speed at baseline - speed at 8 weeks. Higher score indicates better outcome. There are no minimum or maximum values, as this is the measure of the time it takes a participant to walk 25 feet. Higher score indicates higher speed, which is preferable.
Time Frame: Change from baseline to 8 weeks
Population: Only study completers were included in the analysis.
Measure: Mean (Standard Deviation); unit: feet/second
Arm/Group | Time Restricted Feeding
Number analyzed (Participants) | 11
feet/second | -.3 (1.2)
Statistical Analysis 1: Comparison: Time Restricted Feeding; This was a feasibility study and was not powered to detect statistical significance. Significance values are presented but no conclusion of significance can be made; Test type: Other — Single group, within subject pre/post change; p = .39, t-test, 2 sided; Paired-samples t-test

2. Secondary Outcome: Short Form McGill Pain Questionnaire
Description: 15-item questionnaire requiring respondent to rate types of pain as mild, moderate or severe. Scores range from 0-45, with higher pain intensity indicated by higher score. Change calculated as SFMPQ score at basline - SFMPQ score at 8 weeks.
Time Frame: Change from baseline to 8 weeks
Population: Completers only
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Time Restricted Feeding
Number analyzed (Participants) | 11
score on a scale | -1.9 (5.4)
Statistical Analysis 1: Comparison: Time Restricted Feeding; This was a feasibility study and was not powered to detect statistical significance. Significance values are presented but no evaluation of significance can be concluded; Test type: Other — Single group, within subject pre/post change; p = .3, t-test, 2 sided; Paired-samples t-test

3. Secondary Outcome: Modified Fatigue Impact Scale
Description: 21-item questionnaire with possible score ranging from 0-84. Higher scores indicate higher impact of fatigue on a person's life. Change in MFIS was calculated as MFIS score at baseline - MFIS score at 8 weeks.
Time Frame: Change from baseline to 8 weeks
Population: Completers only
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Time Restricted Feeding
Number analyzed (Participants) | 11
score on a scale | -1.3 (14.3)
Statistical Analysis 1: Comparison: Time Restricted Feeding; [analysis description as in outcome 2, analysis 1]; Test type: Other — Single group, within subjects pre/post change; p = .77, t-test, 2 sided; Paired-sample t-test

4. Secondary Outcome: Fatigue Severity Scale
Description: 9-item questionnaire in respondents rate each statement from strongly disagree to strongly agree. Total scores range from 9- 63, with higher score indicating higher fatigue severity. Change in FSS calculated as FSS at baseline - FSS at 8 weeks.
Time Frame: Change from baseline to 8 weeks
Population: Completers only
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Time Restricted Feeding
Number analyzed (Participants) | 11
score on a scale | 2.3 (16.7)
Statistical Analysis 1: Comparison: Time Restricted Feeding; [analysis description as in outcome 2, analysis 1]; Test type: Other — Single group, within subjects pre/post change; p = .66, t-test, 2 sided; Paired-samples t-test

5. Secondary Outcome: Pittsburgh Sleep Quality Index
Description: 19 self-rated items that produce 7 component scores and 1 global score. Only global scores were calculated for this study. Global scores can range from 0-21, with higher scores indicating poorer sleep quality. Change in PSQI calculated as PSQI at baseline - PSQI at 8 weeks.
Time Frame: Change from baseline to 8 weeks
Population: Completers only
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Time Restricted Feeding
Number analyzed (Participants) | 11
score on a scale | .2 (4.0)
Statistical Analysis 1: Comparison: Time Restricted Feeding; [analysis description as in outcome 2, analysis 1]; Test type: Other — Single group, within subjects pre/post change; p = .88, t-test, 2 sided; Paired samples t-test

6. Secondary Outcome: Percent Lean Mass
Description: Lean mass as a percent of total body mass, measured by dual energy x-ray absorptiometry (DXA)
Time Frame: Change from baseline to 8 weeks
Population: Completers only
Measure: Mean (Standard Error); unit: percentage of total mass
Arm/Group | Time Restricted Feeding
Number analyzed (Participants) | 11
percentage of total mass | 0 (1.0)
Statistical Analysis 1: Comparison: Time Restricted Feeding; [analysis description as in outcome 2, analysis 1]; Test type: Other — Single group, within subjects pre/post change; p = .03, t-test, 2 sided; Paired-samples t-test

7. Secondary Outcome: 9 Hole Peg Test Speed
Description: Higher score indicates better outcome. Speed on 9 hole peg test was measured as pegs per second, and change in speed was calculated as speed at baseline - speed at 8 weeks. There are no minimum or maximum values, as the measure is time that it takes a person to complete the test. Higher score indicates faster speed, which is preferable.
Time Frame: Change from baseline to 8 weeks
Population: Completers only
Measure: Mean (Standard Deviation); unit: pegs/second
Arm/Group | Time Restricted Feeding
Number analyzed (Participants) | 11
pegs/second | .02 (.03)
Statistical Analysis 1: Comparison: Time Restricted Feeding; [analysis description as in outcome 2, analysis 1]; Test type: Other — Single group, within subjects pre/post change; p = .06, t-test, 2 sided; Paired samples t-test

8. Secondary Outcome: Symbol Digit Modalities Test (SDMT)
Description: The score is the number of symbols identified correctly in 90 seconds. Potential scores range from 0-110. Higher score indicate improved outcome. Change in score on the SDMT calculated as SDMT score at baseline- SDMT score at 8 weeks.
Time Frame: Change from baseline to 8 weeks
Population: Completers only
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Time Restricted Feeding
Number analyzed (Participants) | 11
score on a scale | 5.8 (8.3)
Statistical Analysis 1: Comparison: Time Restricted Feeding; [analysis description as in outcome 2, analysis 1]; Test type: Other — Single group, within subjects pre/post change; p = .04, t-test, 2 sided; Paired samples t-test

9. Secondary Outcome: Percent Fat Mass
Description: Change in fat mass as percentage of total body mass, measured by DXA. Calculated as percent fat mass at baseline- percent fat mass at 8 weeks.
Time Frame: Change from baseline to 8 weeks
Population: Completers only
Measure: Mean (Standard Deviation); unit: percentage of total mass
Arm/Group | Time Restricted Feeding
Number analyzed (Participants) | 11
percentage of total mass | 0 (1.0)
Statistical Analysis 1: Comparison: Time Restricted Feeding; [analysis description as in outcome 2, analysis 1]; Test type: Other — Single group, within subjects analysis; p = 0, t-test, 2 sided; Paired sample t-test

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Time Restricted Feeding
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

LIMITATIONS AND CAVEATS:
This was a feasibility study and was not powered to detect statistical significance. Significance values are presented but no evaluation of significance can be concluded.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-09-20): https://cdn.clinicaltrials.gov/large-docs/70/NCT04389970/Prot_SAP_ICF_000.pdf